CLINICAL TRIAL: NCT04757623
Title: COMPARISON OF PURSE-STRING CLOSURE VERSUS CONVENTIONAL PRIMARY CLOSURE FOLLOWING STOMA REVERSAL TO REDUCE SURGICAL SITE INFECTION RATE"
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Combined Military Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, Dr Anum Arif, Anum Arif, Combined Military Hospital, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LahoreGeneralHospital
Record Dates: First submitted 2021-02-13; First posted 2021-02-17 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Surgical Site Infection; Difference in Surgical Site Infection According to Gender and Age Groups
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: randomised control trial of two arms
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group B : conventional primary closure (No Intervention): allileostomies are reversed with conventional method
- Group A: Purse string closure (Experimental): the ileostomy reversal circular incision used with stitches of continuous and non-absorbable. The wound of skin was closed by using (Proline No. 1) that leaving 0.5 cm defect on middle in the skin.
  Interventions: Procedure: Purse string closure of Ileostomy

INTERVENTIONS:
Procedure: Purse string closure of Ileostomy — conventional proceedure
  Arms: Group A: Purse string closure

SUMMARY:
The study will be carried out in Surgical Unit-III, Lahore General Hospital, Lahore for one year . . Patients undergoing surgery for Ileostomy will be randomly divided into two groups, Group-A (Purse-string closure) and Group-B (Conventional primary closure). All the patients will be called for follow up checkup on 14th days after operation and after one month. Both of the groups will be checked and recorded for SSI after operation and hospital stay.

DETAILED DESCRIPTION:
The study will be carried out in Surgical Unit-III, Lahore General Hospital. It will be a randomized control trial. Patients undergoing surgery for Ileostomy were randomly divided into two groups, Group-A (Purse-string closure) and Group-B (Conventional primary closure). All the patients will be called for follow-up checkup on 14th days after operation and after one month. Both of the groups will be checked and recorded for SSI after operation and hospital stay. The data will be statistically analyzed by using SPSS v23.0.t test (independent sample) used for the comparison of hospital stay mean. Chi-square will also used for the comparison of the frequencies of SSI. Data were stratified for gender and age. A p-value ≤0.05 will be considered as significant.

ELIGIBILITY:
Inclusion Criteria:

* included in the study 1. Patients of both gender 2. Patients ages between 25-70 3. Patients undergoing surgery for having ileostomy for benign disease of intestine (as per operational definitions).

Exclusion Criteria:

* Following patients were excluded 1. Patients with pre-existing stomal site wound infection 2. Reversal of stoma through laparatomy 3. Post-operative anastomotic leak 4. Ureamic patients 5. Patients on chemotherapy and radiations

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-02-16 (Estimated); Primary Completion 2022-02-16 (Estimated); Study Completion 2022-03-16 (Estimated)

PRIMARY OUTCOMES:
Surgical Site infection | 14th post operative day
  surgical site infection was graded according to southampton score grade IV and V

CONTACTS AND LOCATIONS:
Locations (2):
- Pakistan (2):
  - Anum Arif, Lahore, Select A State Or Province
  - Ammad Asim, Karachi

IPD SHARING:
Plan to Share IPD: No